CLINICAL TRIAL: NCT05638646
Title: A Prospective, Multicentre, Cluster Randomised Controlled Trial to Evaluate the Impact of the Implementation of COPD Quality Standards in High Exacerbation Risk Patients------- A COPD Quality Improvement Program（QIP）
Brief Title: A COPD Quality Improvement Program（QIP）
Acronym: QIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ESR-21-21293
Record Dates: First submitted 2022-11-11; First posted 2022-12-06 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The intervention was delivered at the hospital level. The intervention group will receive QS implementation, including QS training for physicians of respiratory department every 12 weeks; QS implementation check every 12 weeks, and follow-up every 12 weeks, QS-related written COPD clinical procedures will be also suggested to established key QS training requirements are:1) COPD diagnosis and assessment; 2)Therapy prescribed in accordance with national guideline 3)Non-pharmacological interventions; 4)An appropriate follow-up according to QS.
  The control group will maintain current practice and follow up every 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): Practice standard for clinical diagnosis and treatment of chronic obstructive pulmonary disease
  Interventions: Other: Intervention group
- control group (Other): Maintain current treatment
  Interventions: Other: control group

INTERVENTIONS:
Other: Intervention group — Practice standard for clinical diagnosis and treatment of chronic obstructive pulmonary disease
  Arms: Intervention group
Other: control group — Maintain current treatment
  Arms: control group

SUMMARY:
QIP(Quality Improvement Programme) is a COPD quality improvement program in China. The initial step of this program is to set up the Quality Standards(QS) of COPD management in clinical practice, then embed Quality Standards into routine care and uses Quality Control Indicators (QCI)to check the QS implementation. The aim of the QIP program is to standardize COPD management in clinical practice in China, including the standardization of diagnosis, assessment, pharmacological and non-pharmacological intervention, and follow-up. COPD patients can benefit from standardization clinical behaviours, to be identified early, be accessed comprehensively, and be treated correctly according to guidelines, and with an appropriate follow-up to improve adherence.

DETAILED DESCRIPTION:
Background and Rationale Chronic obstructive pulmonary disease (COPD) is currently the most common chronic respiratory disease in China which causes a huge economic and social burden. Acute Exacerbation is a crucial issue that cannot be ignored in the management of COPD. Patients with frequent exacerbations have been found to have greater airflow limitation, a greater symptom burden, increased mortality, and worsen the quality of life (QoL). However, The COPD management of those patients in clinical practice is poor in China. Patients with a low standard of care, lack of regularly pharmacological and non-pharmacological intervention, and insufficient follow-up and disease education in clinical practice.

Objectives and Outcomes QIP(Quality Improvement Programme) is a COPD quality improvement program in China. The initial step of this program is to set up the Quality Standards(QS) of COPD management in clinical practice, then embed Quality Standards into routine care and uses Quality Control Indicators (QCI)to check the QS implementation. The aim of the QIP program is to standardize COPD management in clinical practice in China, including the standardization of diagnosis, assessment, pharmacological and non-pharmacological intervention, and follow-up. COPD patients can benefit from standardization clinical behaviours, to be identified early, be accessed comprehensively, and be treated correctly according to guidelines, and with an appropriate follow-up to improve adherence.

The objective of QIP study is to address key gaps in management of patients with high-risk through a targeted quality improvement programme in a healthcare system or practice. The aim is to evaluate the impact of QS implementation on target population compared to usual care in a real-world setting, including but not limited to COPD exacerbation, lung function, quality of life, and treatment pattern.

Study design This is a interventional, cluster-randomized, pragmatic clinical study. A total of 41 hospitals will be selected. Among them, 40 eligible hospitals will be selected across China and randomized (stratified by tier and geographic region) to the intervention group or control group at the ratio of 1:1. In addition, the leading site will be assigned to the intervention group without following the randomization procedure. In the intervention group, QS implementation will be performed. The control group will maintain the current practice. Eligible patients will be recruited in both groups and will be followed up every 12 weeks for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with COPD
2. Aged 40 years or older
3. CAT≥10
4. With exacerbation history：

   1. at least 2 moderate or 1 severe exacerbation in the previous year
   2. or 1 moderate exacerbation in the previous year with FEV1 <50% predicted value at baseline;
5. Must able to sign the informed consent form

Exclusion Criteria:

1. Patients on triple therapy at baseline with a LAMA, LABA, and inhaled corticosteroid (ICS) combination (Including open triple and fix-dose triple)
2. Significant diseases or conditions other than COPD, which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study
3. Patients who are currently involved in any other interventional studies

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1107 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to clinically important deterioration (CID) | 48 weeks
  Time to CID, which is defined as the time from the date of enrolment until the date of the first CID.CID defined as any of the following events:1) Trough FEV1 decline ≥100ml;2) CAT increasing ≥ 2 unit;3) one moderate or severe exacerbation.

SECONDARY OUTCOMES:
Annual rate of moderate or severe COPD exacerbation | 1 year
  Annual rate of moderate or severe COPD exacerbation
Annual rate of severe COPD exacerbation | 1 year
  Annual rate of severe COPD exacerbation
Change from baseline in trough FEV1 over 48 weeks | 48 weeks
  Change from baseline in trough FEV1 over 48 weeks
Change from baseline in CAT over 48 weeks | 48 weeks
  Change from baseline in CAT over 48 weeks
Proportion of patients received inhalation technique review at least once during follow-up period | 48 weeks
  Proportion of patients received inhalation technique review at least once during follow-up period
Proportion of patients received long-acting inhaled medicine with percentage of days covered (PDC)≥ 80% over 48 weeks | 48 weeks
  Proportion of patients received long-acting inhaled medicine with percentage of days covered (PDC)≥ 80% over 48 weeks
Proportion of prescription of inhaled maintenance medicine at 12 weeks | 12 weeks
  Proportion of prescription of inhaled maintenance medicine at 12 weeks
Proportion of prescription of inhaled maintenance medicine at 24 weeks | 24 weeks
  Proportion of prescription of inhaled maintenance medicine at 24 weeks
Proportion of prescription of inhaled maintenance medicine at 36 weeks | 36 weeks
  Proportion of prescription of inhaled maintenance medicine at 36 weeks
Proportion of prescription of inhaled maintenance medicine at 48 weeks | 48 weeks
  Proportion of prescription of inhaled maintenance medicine at 48 weeks
Proportion of patients prescribed ICS-containing inhaled maintenance medicine at 12 weeks | 12 weeks
  Proportion of patients prescribed ICS-containing inhaled maintenance medicine at 12 weeks
Proportion of patients prescribed ICS-containing inhaled maintenance medicine at 24 weeks | 24 weeks
  Proportion of patients prescribed ICS-containing inhaled maintenance medicine at 24 weeks
Proportion of patients prescribed ICS-containing inhaled maintenance medicine at 36 weeks | 36 weeks
  Proportion of patients prescribed ICS-containing inhaled maintenance medicine at 36 weeks
Proportion of patients prescribed ICS-containing inhaled maintenance medicine at 48 week | 48 weeks
  Proportion of patients prescribed ICS-containing inhaled maintenance medicine at 48 week

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, Professor, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

DOCUMENTS (1):
  • Study Protocol (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT05638646/Prot_000.pdf